CLINICAL TRIAL: NCT05691127
Title: Burden of Respiratory Illnesses in Pediatric Intensive Care Unit and Its Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hadier Khaled Mahmoud, resident at pediatric departement at el helal hospital, Sohag University
Other Study IDs: soh-Med-22-12-08
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Respiratory Illnesses
MeSH Terms: interventions — Blood Cell Count; Diagnostic Imaging; Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Respiratory Diseased children
  Interventions: Diagnostic Test: Complete blood count (CBC), C reactive protein (CRP(., Chest x ray, ABG, Electrolytes, Random blood sugar, Creatinine

INTERVENTIONS:
Diagnostic Test: Complete blood count (CBC), C reactive protein (CRP(., Chest x ray, ABG, Electrolytes, Random blood sugar, Creatinine — I will use these investigations in my study

SUMMARY:
Acute respiratory infections (ARI) are an important cause of mortality and morbidity among children; one-fifths of under-five mortality being contributed by them (predominantly pneumonias ).

About 11.9 million episodes of severe and 3.0 million episodes of very severe acute lower respiratory infections (ALRI) result in hospital admissions in young children worldwide.

Respiratory infections and illnesses in children thus form a substantial disease burden in Pediatric intensive care unit. With this is mind, we studied clinical profile and risk factors contributing to mortality, and outcome of children with acute respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

Children with pneumonia, bronchiolitis, bronchial asthma, chemical pneumonitis, cystic fibrosis and other respiratory diseases, Cardiorespiratory cases and Neurological cases with respiratory illness

Exclusion Criteria:

Post trauma case. Postoperative cases (developing respiratory complications during PICU stay).

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with pneumonia, bronchiolitis, bronchial asthma, chemical pneumonitis, cystic fibrosis and other respiratory diseases, Cardiorespiratory cases and Neurological cases with respiratory illness
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
incidence of respiratory illnesses | one year
  incidence of respiratory illnesses in PICU among other children

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khilnani P, Sarma D, Singh R, Uttam R, Rajdev S, Makkar A, Kaur J. Demographic profile and outcome analysis of a tertiary level pediatric intensive care unit. Indian J Pediatr. 2004 Jul;71(7):587-91. doi: 10.1007/BF02724117. PMID 15280607
- [Background] Nair H, Simoes EA, Rudan I, Gessner BD, Azziz-Baumgartner E, Zhang JSF, Feikin DR, Mackenzie GA, Moiisi JC, Roca A, Baggett HC, Zaman SM, Singleton RJ, Lucero MG, Chandran A, Gentile A, Cohen C, Krishnan A, Bhutta ZA, Arguedas A, Clara AW, Andrade AL, Ope M, Ruvinsky RO, Hortal M, McCracken JP, Madhi SA, Bruce N, Qazi SA, Morris SS, El Arifeen S, Weber MW, Scott JAG, Brooks WA, Breiman RF, Campbell H; Severe Acute Lower Respiratory Infections Working Group. Global and regional burden of hospital admissions for severe acute lower respiratory infections in young children in 2010: a systematic analysis. Lancet. 2013 Apr 20;381(9875):1380-1390. doi: 10.1016/S0140-6736(12)61901-1. Epub 2013 Jan 29. PMID 23369797
- [Background] Tan GH, Tan TH, Goh DY, Yap HK. Risk factors for predicting mortality in a paediatric intensive care unit. Ann Acad Med Singap. 1998 Nov;27(6):813-8. PMID 10101556